CLINICAL TRIAL: NCT00354861
Title: A Phase I, Single-Blind Study to Determine the Safety, Tolerability and Pharmacodynamic Profiles of a Hepatitis B Antigen Combined With IMP321 Versus the Hepatitis B Antigen Alone and a Reference Vaccine in Healthy Young Male Volunteers
Brief Title: A Randomized Phase I Study of a Hepatitis B Antigen Combined With IMP321
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immutep S.A.S. (Industry)
Collaborators: SGS Aster-Cephac (CRO) (Unknown)
Responsible Party: F. Triebel, Chief Medical Officer, Immutep S.A.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: P002; Aster-P020256
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2008-04-25 (Estimated); Status verified 2008-04

CONDITIONS: Healthy
Keywords: Healthy volunteers; IMP321; Adjuvant; Pharmacodynamics
MeSH Terms: interventions — Hepatitis B Antigens; Engerix-B

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): IMP321
  Interventions: Biological: hepatitis B antigen (without alum) plus IMP321
- B (Placebo Comparator): Saline
  Interventions: Biological: hepatitis B antigen alone (without alum)
- C (Active Comparator): Engerix B
  Interventions: Biological: Engerix B

INTERVENTIONS:
Biological: hepatitis B antigen (without alum) plus IMP321 — hepatitis B antigen (10 µg HbsAg, subtype adw, without alum) with IMP321
  Other Names: CD223; hLAG-3Ig; LAG-3
  Arms: A
Biological: hepatitis B antigen alone (without alum) — hepatitis B antigen (10 µg HbsAg, subtype adw, without alum) with physiological saline
  Arms: B
Biological: Engerix B — 20 µg hepatitis B antigen absorbed on alum
  Arms: C

SUMMARY:
This is a single centre, three single administrations (Days 1, 29 and 57) at increasing doses of IMP321 (3, 10, 30 and 100 µg) in four cohorts of 12 subjects, single blind, randomized study.

DETAILED DESCRIPTION:
In each cohort, 8 subjects will receive the hepatitis B antigen (10 µg) with IMP321 at one dose, 2 subjects will receive the reference hepatitis B antigen (10 µg) alone with physiological saline and 2 subjects will receive the commercial vaccine Engerix B® (20 µg).

Engerix B® will be administered intramuscularly. The other treatments will be administered subcutaneously.

The four successive cohorts of volunteers will be:

Cohort A:

* 8 subjects treated by hepatitis B antigen (10 µg HbsAg, subtype adw, without alum) with IMP321 (3 µg),
* 2 subjects treated by hepatitis B antigen (10 µg HbsAg, subtype adw, without alum) with physiological saline,
* 2 subjects treated by the commercial hepatitis vaccine Engerix B® (20 µg HBsAg with alum).

If the tolerability of this cohort is acceptable, the following cohort will be done.

Cohort B:

* 8 subjects treated by hepatitis B antigen (10 µg HbsAg, subtype adw, without alum) with IMP321 (10 µg),
* 2 subjects treated by hepatitis B antigen (10 µg HbsAg, subtype adw, without alum) with Physiological saline,
* 2 subjects treated by the commercial hepatitis vaccine Engerix B® (20 µg HBsAg with alum).

If the tolerability of this cohort is acceptable, the following cohort will be done.

Cohort C:

* 8 subjects treated by hepatitis B antigen (10 µg HbsAg, subtype adw, without alum) with IMP321 (30 µg),
* 2 subjects treated by hepatitis B antigen (10 µg HbsAg, subtype adw, without alum) with physiological saline,
* 2 subjects treated by the commercial hepatitis vaccine Engerix B® (20 µg HBsAg with alum).

If the tolerability of this cohort is acceptable, the following cohort will be done.

Cohort D:

* 8 subjects treated by hepatitis B antigen (10 µg HbsAg, subtype adw, without alum) with IMP321 (100 µg),
* 2 subjects treated by hepatitis B antigen (10 µg HbsAg, subtype adw, without alum) with physiological saline
* 2 subjects treated by the commercial hepatitis vaccine Engerix B® (20 µg HBsAg with alum).

Blood samples will be collected on the morning of days 1, 29, 36, 57 and 85 for pharmacodynamic evaluation.

Monitoring for the occurrence of adverse events (AE), changes in physical examination, vital signs (blood pressure, pulse rate, respiration), electrocardiograms (ECG) and clinical laboratory tests (biochemistry, haematology, urinalysis) will be performed before and after each dose of the study drug to assess safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* able to give a written informed consent ;
* healthy male volunteers aged between 18 and 40 years and post-menopausal healthy women aged between 18 and 55 years;
* with body mass index (weight/height²) in the range 18 to 30 kg/m²;
* registered with the French Social Security in agreement with the French Law (Huriet Law : N° 88.1138 - 20.12.88) on biomedical experimentation;
* able to comply with protocol requirements, including overnight stays, blood and urine sample collections as defined in the protocol;
* not previously vaccinated for Hepatitis B.

Exclusion Criteria:

* who on direct questioning and physical examination have evidence of any clinically significant acute or chronic disease, including known or suspected HIV, HBV and HCV infection ;
* with any clinically significant abnormality following review of pre-study laboratory tests and full physical examination ;
* who have received any experimental drug within the exclusion period defined in the National Register for Healthy Volunteers of the French Ministry of Health ;
* who forfeit their freedom by administrative or legal award or who were under guardianship ;
* unwilling to give their informed consent ;
* who present a positive laboratory test for Hepatitis B surface antigen (HbsAg), HBc antibodies, HIV 1 and 2 antibodies and HCV antibodies ;
* who have a history of allergy or intolerance to the study drug ;
* who had a history of serious allergy, asthma, allergic skin rash or sensitivity to any drug ;
* who are known or suspected alcohol or drug abusers ;
* who present a positive laboratory test for urine drug screening (opiates, barbiturates, amphetamine, cannabis) ;
* who undergo surgery or have donated blood within 1 month prior to the start of the study ;
* who have taken any prescribed or over the counter drug (including antacid drug), with the exception of paracetamol (up to 3 g per day) within 1 week prior to the first dose administration ;
* who receive any drug known to affect hepatic metabolism like cimetidine, ketoconazole, fluconazole, itraconazole, phenytoin, rifampicin, rifabutin within 1 month prior to the first dose administration ;
* who receive any drug known to affect renal tubular secretion like probenecid, beta-lactam antibiotics within 2 weeks prior to the first dose administration ;
* who present any clinical condition or prior therapy which, in the opinion of the investigator, made the subject unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2005-05; Primary Completion 2005-11 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
To evaluate clinical and laboratory safety and tolerability profiles | 3 months

SECONDARY OUTCOMES:
To determine T cell response induction efficacy | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Didier Chassard, M.D., Principal Investigator — SGS Aster-Cephac
Locations (1):
- SGS Aster-Cephac, Paris, France

REFERENCES:
- See also: Sponsor's website — http://www.immutep.com